CLINICAL TRIAL: NCT00863746
Title: A Phase III, Multi-center, Placebo-Controlled Trial of Sorafenib (BAY43-9006) in Patients With Relapsed or Refractory Advanced Predominantly Non Squamous Non-Small Cell Lung Cancer (NSCLC) After 2 or 3 Previous Treatment Regimens for Advanced Disease
Brief Title: A 3rd/4th Line Placebo-controlled Trial of Sorafenib in Patients With Predominantly Non Squamous Non-Small Cell Lung Cancer (NSCLC).
Acronym: MISSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13266; 2008-006914-62 (EudraCT Number)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma; Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer (NSCLC); Sorafenib
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Participants received 2 tablets of Sorafenib (2×200 mg) orally twice daily (BID)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Participants received 2 tablets of placebo orally twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg twice daily (BID)
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Placebo - 2 tablets twice daily (BID)
  Arms: Placebo

SUMMARY:
The purpose of the study is to see if sorafenib plus best supportive care (i.e. in addition to the non-cancer treatments patients would normally receive) is an effective treatment for lung cancer compared to best supportive care alone. The safety and tolerability of the two treatment groups will also be compared. The goal of the study is to test the ability of sorafenib to improve survival compared to best supportive care alone.

DETAILED DESCRIPTION:
Acronyms used in Adverse Events section: Disseminated intravascular coagulation (DIC), International normalized ratio (INR), Atrioventricular (AV), Gastrointestinal (GI), Not otherwise specified (NOS), Common Terminology Criteria for Adverse Events (CTCAE), Absolute neutrophil count (ANC), Central nervous system (CNS), Acute respiratory distress syndrome (ARDS), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written Informed Consent
* Advanced relapsed or refractory predominantly non squamous NSCLC. The diagnosis must have been confirmed cyto-/ histologically
* Patients must have measurable or non-measurable disease
* At least two but not more than three prior standard treatment regimens for NSCLC
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Male or female subjects >/= 18 years of age (>/=20 for Japan) at the time of Informed Consent
* Life expectancy of at least 12 weeks
* Ability to swallow oral medication
* Both men and women using adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of the study drug:

  * Haemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) >1,500/mm3
  * Platelet count >/= 100,000/µl
  * Total bilirubin </=1.5 x the upper limit of normal
  * Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (</= 5 x upper limit of normal in patients with liver metastases) Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (</= 5 x upper limit of normal in patients with liver metastases)
  * Alkaline phosphatase < 4 x upper limit of normal (</= 5 x upper limit of normal in patients with liver metastases)
  * Prothrombin Time (PT)-International Normalized Ratio (INR) or Partial Thromboplastin Time (PTT) < 1.5 x upper limit of normal
  * Serum creatinine < 1.5 x upper limit of normal
  * Calculated creatinine clearance of >/= 50 mL/min

Exclusion Criteria:

* NSCLC patients with predominantly squamous cell carcinoma histology

Excluded medical conditions:

* History of cardiac disease: Congestive heart failure, Active coronary artery disease (CAD), Cardiac arrhythmias (>Grade 2 NCI-CTCAE [National Cancer Institute-Common Terminology Criteria for Adverse Events] vers. 3.0)
* Uncontrolled hypertension despite two anti-hypertensive medications
* History of Human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* History of organ allograft
* Active clinically serious infections (> grade 2 NCI-CTCAE vers. 3.0)
* Patients with seizure disorder requiring medication
* Patients with evidence or history of bleeding diathesis or coagulopathy
* Patients undergoing renal dialysis
* Pulmonary hemorrhage/ bleeding event >/= CTCAE grade 2 within four weeks prior to the first dose of the study drug
* Any other hemorrhage/ bleeding event >/= CTCAE grade 3 within four weeks prior to the first dose of the study drug
* Thrombotic or embolic venous or arterial events such as cerebrovascular accident
* Pregnant or breast-feeding women.
* Any condition which could affect the absorption or pharmacokinetics of the study drug
* Prior treatment with other Vascular Endothelial Growth Factor (VEGF) (R) inhibitors, including compounds that impact vascularity (i.e. sunitinib, thalidomide, vandetanib, vascular disrupting agents [VDA], VEGF-trap and other experimental agents of this class). Only bevacizumab (Avastin) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (157):
- United States (3):
  - Fayetteville, Arkansas
  - Stanford, California
  - Philadelphia, Pennsylvania
- Argentina (5):
  - Ramos Mejía, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - Santa Fé
- Austria (3):
  - Vienna, Vienna
  - Graz
  - Linz
- Belgium (4):
  - Antwerp
  - Bruxelles - Brussel
  - Charleroi
  - Genk
- Brazil (6):
  - Brasília, Federal District
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São José dos Campos, São Paulo
  - São Paulo, São Paulo
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Montreal, Quebec, Canada
- Chile (2):
  - Santiago, Santiago Metropolitan
  - Santiago
- China (7):
  - Guangzhou, Guangdong
  - Nanjing, Jiangsu
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Guangzhou
  - Shanghai
- France (8):
  - Caen
  - Dijon
  - La Roche-sur-Yon
  - La Tronche
  - Lille
  - Lyon
  - Saint-Herblain
  - Tours
- Germany (11):
  - Heidelberg, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Gauting, Bavaria
  - München, Bavaria
  - Hamburg, Hamburg
  - Kassel, Hesse
  - Cologne, North Rhine-Westphalia
  - Großhansdorf, Schleswig-Holstein
  - Bad Berka, Thuringia
- Greece (3):
  - Athens
  - Heraklion
  - Thessaloniki
- Hong Kong (3):
  - Shatin, N.T
  - Hong Kong
  - Kowloon
- Hungary (5):
  - Budapest
  - Edelény
  - Farkasgyepű
  - Törökbálint
  - Zalaegerszeg
- India (3):
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Kerala
- Indonesia (2):
  - Bandung
  - Jakarta
- Israel (5):
  - Zrifin, Israel
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
- Italy (9):
  - Rozzano, Milano
  - Monza, Monza-Brianza
  - Orbassano, Torino
  - Avellino
  - Genova
  - Livorno
  - Parma
  - Perugia
  - Roma
- Japan (8):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Fukuoka, Fukuoka
  - Akashi, Hyōgo
  - Sakai, Osaka
  - Sayama, Osaka
  - Itabashi-ku, Tokyo
  - Koto-ku, Tokyo
- Netherlands (6):
  - Amsterdam
  - Harderwijk
  - Heerlen
  - Helmond
  - Nieuwegein
  - Zwolle
- Pakistan (2):
  - Lahore, Punjab Province
  - Karachi, Sindh
- Peru (3):
  - Callao
  - Lima
  - San Borja
- Philippines (4):
  - Cebu City
  - Manila
  - Metro Manila
  - Quezon City
- Poland (6):
  - Kielce
  - Krakow
  - Olsztyn
  - Rzeszów
  - Szczecin
  - Warsaw
- Russia (4):
  - Kazan'
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Singapore, Singapore
- South Africa (5):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Prietoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- South Korea (2):
  - Seoul, Seoul Teugbyeolsi
  - Seoul
- Spain (9):
  - Barcelona, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Lleida, Lleida
  - Lugo, Lugo
  - Madrid, Madrid
  - Málaga, Málaga
  - Ourense, Ourense
  - Seville, Sevilla
  - Zamora, Zamora
- Sweden (5):
  - Falun
  - Gothenburg
  - Linköping
  - Lund
  - Stockholm
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla
- Turkey (Türkiye) (5):
  - Ankara
  - Instanbul
  - Istanbul
  - Izmir
  - Kocaeli
- United Kingdom (7):
  - Bristol, Avon
  - Cambridge, Cambridgeshire
  - London, London
  - Greater Manchester, Manchester
  - Sutton, Surrey
  - Leeds, West Yorkshire
  - Aberdeen

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 350 | 353
Participants Received Treatment | 346 (Safety population) | 351 (Safety population)
Completed | 279 | 318
Not Completed | 71 | 35
Not completed — Not treated | 4 | 2
Not completed — Adverse Event | 41 | 16
Not completed — non-compliant with study medication | 4 | 0
Not completed — Consent withdrawn | 15 | 14
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 5 | 3
Not completed — Other | 1 | 0
Period: Survival Follow up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 298 (298 patients of 317 patients (= 346 randomized - 29 deaths) entered the survival follow-up) | 331 (331 patients of 339 patients (=353 randomized - 14 death) entered the survival follow-up.)
Completed | 45 | 51
Not Completed | 253 | 280
Not completed — Death | 244 | 271
Not completed — Lost to Follow-up | 2 | 1
Not completed — Consent Withdrawn | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 350 | 353 | 703
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (10.7) | 60.9 (9.8) | 59.9 (10.3)
Age, Customized [Number; unit: Participants]
  < 65 years | 239 | 222 | 461
  >= 65 and < 75 years | 91 | 102 | 193
  >= 75 years | 20 | 29 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 144 | 308
  Male | 186 | 209 | 395
Region (CRF [case report form]) [Number; unit: Participants]
  Group 1 (North America, Northern/Western Europe) | 122 | 119 | 241
  Group 2 (S. America, Eastern Europe, Asia-Pacific) | 228 | 234 | 462
Number of participants with prior anti-cancer therapy and diagnostic procedures [Number; unit: Participants]
  2 regimens | 188 | 197 | 385
  3 regimens | 158 | 153 | 311
  4 regimens | 3 | 3 | 6
  5 regimens | 1 | 0 | 1
Brain metastasis [Number; unit: Participants]
  No | 293 | 299 | 592
  Yes | 56 | 54 | 110
  Missing | 1 | 0 | 1
Prior EGFR (Epidermal Growth Factor Receptor) inhibitor treatment [Number; unit: Participants]
  No | 141 | 146 | 287
  Yes | 209 | 207 | 416
ECOG (Eastern Cooperative Oncology Group) performance status [Number; unit: Participants] — A scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst).
  Participants
    Missing | 6 | 1 | 7
    0 | 110 | 110 | 220
    1 | 233 | 242 | 475
    2 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from date of randomization to date of death due to any cause. Overall survival of subjects alive at the time of analysis will be censored at their last date of follow-up or database cut off date whichever came first.
Time Frame: From randomization of the first subject until 36 months later
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 350 | 353
Days | 248 [224 to 290] | 253 [231 to 301]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test for superiority of Sorafenib over Placebo; Test type: Superiority or Other; p = 0.4687, Log Rank — p-value of one-sided test (significance level 2.5%); stratified by region, number of prior treatments, presence brain mets at baseline, prior EGFR inhibitor treatment; Hazard Ratio (HR) = 0.9934, 95% CI 2-sided [0.8409 to 1.1735]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from date of randomization to date of first observed disease progression (radiological or clinical, whichever is earlier) or death due to any cause, if death occurs before progression is documented. Progressive Disease (PD) is defined as at least a 20% increase in the sum of longest diameter (LD) of measured lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Appearance of new lesions will also constitute progressive disease. In exceptional circumstances unequivocal progression of a non-measured lesion may be accepted as evidence of disease progression.
Time Frame: From randomization of the first subject until 36 months later assessed every 6 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 350 | 353
Days | 84 [81 to 86] | 43 [42 to 44]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test for superiority of Sorafenib over Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — p-value of one-sided test (significance level 2.5%); stratified by region, number of prior treatments, presence brain mets at baseline, prior EGFR inhibitor treatment; Hazard Ratio (HR) = 0.6068, 95% CI 2-sided [0.5139 to 0.7165]

3. Secondary Outcome: Disease Control
Description: Disease control (DC) was defined as the proportion of patients whose best response was Complete Response [CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target)] or Partial Response [PR: at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD] or Stable Disease [SD: steady state of disease which was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD)].
Time Frame: From randomization of the first subject until 36 months later assessed every 6 weeks
Population: Full Analysis Set (FAS)
Measure: Number; unit: Proportion of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 350 | 353
Proportion of participants | 0.4714 | 0.2465
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p < 0.000001, Cochran-Mantel-Haenszel; stratified by region, number of prior treatments, presence brain mets at baseline, prior EGFR inhibitor treatment; CMH-adjusted difference in proportions = 0.2263, 95% CI 2-sided [0.1575 to 0.2952]

4. Secondary Outcome: Objective Tumor Response
Description: Objective tumor response was defined as the proportion of patients whose best response was Complete Response [CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target)] or Partial Response [PR: at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD] over the whole duration of study.
Time Frame: From randomization of the first subject until 36 months later assessed every 6 weeks
Population: Full Analysis Set (FAS)
Measure: Number; unit: Proportion of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 350 | 353
Proportion of participants | 0.0486 | 0.0085
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.000876, Cochran-Mantel-Haenszel; stratified by region, number of prior treatments, presence brain mets at baseline, prior EGFR inhibitor treatment; CMH-adjusted difference in proportions = 0.0390, 95% CI 2-sided [0.0137 to 0.0642]

5. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the time from date of randomization to date of first observed disease progression (radiological or clinical, whichever is earlier).
Time Frame: From randomization of the first subject until 36 months later assessed every 6 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 350 | 353
Days | 89 [84 to 124] | 43 [42 to 44]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test for superiority of Sorafenib over Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — p-value of one-sided test (significance level 2.5%); stratified by region, number of prior treatments, presence brain mets at baseline, prior EGFR inhibitor treatment; Hazard Ratio (HR) = 0.5420, 95% CI 2-sided [0.4526 to 0.6492]

6. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire for Palliative Care (EORTC QLQ-C15-PAL) - Global Health Status
Description: The EORTC QLQ-C15-PAL is an abbreviated 15-item version of the EORTC core quality of life questionnaire (EORTC QLQ-C30) developed for use in palliative care. The 'Global Health status' subscale consists of question 15 of the questionnaire. The score of 'Global Health status' ranges from 0 (very poor) to 100 (excellent). The change of score ranges from -100 (maximum degree of worsening) to 100 (maximum degree of improvement).
Time Frame: Baseline and up to End of treatment (up to Cycle 41, 21 days per cycle)
Population: Patient report outcomes (PRO) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 318 | 332
Scores on a scale
  Cycle 2 (n=295, 309) | -6.158 (22.435) | -3.398 (18.370)
  Cycle 3 (n=233, 188) | -5.222 (19.881) | -2.305 (18.976)
  Cycle 4 (n= 187, 119) | -2.763 (19.700) | -3.782 (16.728)
  Cycle 5 (n= 158, 92) | -3.586 (18.843) | -3.080 (18.806)
  Cycle 6 (n=136, 60) | -5.270 (19.845) | -3.056 (16.089)
  End of treatment (up to Cycle 41, n=192, 221) | -12.153 (24.535) | -12.142 (21.780)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.3121, Mixed Models Analysis — p-value for test of treatment effect equal to 0

7. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) - Coughing Subscale
Description: A clinically valid 13-item tool for assessing disease- and treatment-specific symptoms in lung cancer patients in clinical trials. The coughing subscale uses question 1 of the questionnaire. The scale ranges from 0 to 100. Higher score means higher level of symptomatology/problems. The change of score ranges from -100 (decrease in level of symptomatology/problems) to 100 (increase in level of symptomatology/problems).
Time Frame: Baseline and up to End of treatment (up to Cycle 41, 21 days per cycle)
Population: Patient report outcomes (PRO) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 318 | 332
Scores on a scale
  Cycle 2 (n=297, 314 | 0.786 (25.910) | 2.866 (24.325)
  Cycle 3 (n=234, 192) | -1.567 (24.753) | -0.174 (23.754)
  Cycle 4 (n=187, 121) | -2.674 (26.751) | 0.000 (26.527)
  Cycle 5 (n=154, 92) | -0.216 (25.422) | -1.812 (24.392)
  Cycle 6 (n=134, 61) | -2.239 (23.904) | -3.825 (29.875)
  End of treatment (up to Cycle 41) (n=194, 225) | 8.763 (27.103) | 5.333 (29.734)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.2948, Mixed Models Analysis — p-value for test of treatment effect equal to 0

8. Secondary Outcome: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) - Dyspnea
Description: A clinically valid 13-item tool for assessing disease- and treatment-specific symptoms in lung cancer patients in clinical trials. The dyspnea subscale uses questions 3, 4 and 5 of the questionnaire. The scale ranges from 0 to 100. Higher score means higher level of symptomatology/problems. The change of score ranges from -100 (decrease in level of symptomatology/problems) to 100 (increase in level of symptomatology/problems).
Time Frame: Baseline and up to End of treatment (up to Cycle 41, 21 days per cycle)
Population: Patient report outcomes (PRO) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 318 | 332
Scores on a scale
  Cycle 2 (n=290, 309) | 3.678 (16.251) | 3.740 (17.806)
  Cycle 3 (n=232, 189) | 0.958 (16.021) | 2.058 (17.984)
  Cycle 4 (n=186, 120) | 3.226 (17.258) | 2.963 (16.343)
  Cycle 5 (n=153, 91) | 3.486 (17.169) | 3.419 (17.739)
  Cycle 6 (n=133, 61) | 2.840 (16.843) | 2.004 (14.700)
  End of treatment (up to Cycle 31, n=191, 222) | 12.158 (21.694) | 10.611 (22.738)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.8344, Mixed Models Analysis — p-value for test of treatment effect equal to 0

9. Secondary Outcome: Mean Change From Baseline in EuroQol-5D (EQ-5D) - Index Score
Description: The Euro-Qol 5D (EQ-5D) is a validated assessment tool of Health Related Quality of Life (HRQOL) and utilities consisting of 15 statements. Patients select those statements that best describe their current health state regarding mobility, self-care, usual activities, pain/discomfort, and anxiety/depression which is converted into a utility value. Range of scale is from -0.594 (worst possible health state) to 1 (perfect health) based on UK weights. The change of score ranges from -1.594 (high degree of worsening) to 1.594 (high degree of improvement).
Time Frame: Baseline and up to End of treatment (up to Cycle 41, 21 days per cycle)
Population: Patient report outcomes (PRO) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 318 | 332
Scores on a scale
  Cycle 3 (n=228, 186) | -0.0627 (0.2402) | -0.0386 (0.1998)
  Cycle 5 (n=150, 91) | -0.0439 (0.2022) | -0.0728 (0.2373)
  End of treatment (up to cycle 41) (n=188, 219) | -0.1845 (0.3348) | -0.1442 (0.3108)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.1438, Mixed Models Analysis — p-value for test of treatment effect equal to 0

10. Secondary Outcome: Mean Change From Baseline in EuroQol-5D (EQ-5D) - VAS Score
Description: A visual analogue scale (EQ VAS) used by patients to rate their current health state from 100 (best imaginable health state) to 0 (worst imaginable health state). The change of score ranges from -100 (high degree of worsening) to 100 (high degree of improvement)
Time Frame: Baseline and up to End of treatment (up to Cycle 41, 21 days per cycle)
Population: Patient report outcomes (PRO) analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 318 | 332
Scores on a scale
  Cycle 3 (n=218 , 183) | -3.73 (16.53) | -3.48 (17.35)
  Cycle 5 (n=144, 89) | -5.39 (16.66) | -2.48 (16.37)
  End of treatment (up to Cycle 41, n=184, 216) | -12.72 (16.65) | -10.75 (18.90)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.9228, Mixed Models Analysis — p-value for treatment effect equal to 0

ADVERSE EVENTS:
Groups:
- Sorafenib (Nexavar, BAY43-9006): Participants received 2 tablets of Sorafenib (2x200 mg) orally twice daily (BID)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Serious Adverse Events (participants affected / at risk) | 136/346 | 111/351
Other Adverse Events (participants affected / at risk) | 332/346 | 289/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=346) | Placebo (N=351)
DIC (Blood and lymphatic system disorders) | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
INR (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 2 | 1
Cardiac general - Other (Cardiac disorders) | 2 | 1
Cardiac ischemia/infarction (Cardiac disorders) | 3 | 1
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0
Conduction abnormality, AV Block - 3rd Degree (Complete AV Block) (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular arrhythmia, Atrial Tach/Paroxysmal AT (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 2 | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 0
Ocular - Other (Eye disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 3 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
GI - Other (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 0 | 1
Stricture, GI, Biliary tree (Gastrointestinal disorders) | 0 | 1
Stricture, GI, Esophagus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Constitutional symptoms - Other (General disorders) | 10 | 4
Death not associated with CTCAE term, Death NOS (General disorders) | 2 | 0
Death not associated with CTCAE term, Disease progression NOS (General disorders) | 20 | 13
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 4 | 1
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 1 | 1
Pain, Abdomen NOS (General disorders) | 2 | 2
Pain, Back (General disorders) | 1 | 3
Pain, Bone (General disorders) | 2 | 4
Pain, Chest wall (General disorders) | 2 | 3
Pain, Chest/Thorax NOS (General disorders) | 3 | 2
Pain, Extremity - limb (General disorders) | 0 | 2
Pain, Pain NOS (General disorders) | 1 | 0
Pain, Tumor pain (General disorders) | 1 | 1
Weight loss (General disorders) | 1 | 0
Hepatobiliary - Other (Hepatobiliary disorders) | 1 | 1
Liver dysfunction (Hepatobiliary disorders) | 2 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Infection (Documented clinically), Lung (Pneumonia) (Infections and infestations) | 1 | 1
Infection - Other (Infections and infestations) | 1 | 1
Infection with normal ANC, Bone (Osteomyelitis) (Infections and infestations) | 1 | 0
Infection with normal ANC, Brain (Encephalitis, infectious) (Infections and infestations) | 1 | 0
Infection with normal ANC, Bronchus (Infections and infestations) | 3 | 2
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 11 | 4
Infection with normal ANC, Skin (cellulitis) (Infections and infestations) | 1 | 0
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 2 | 1
Infection with unknown ANC, Lung (Pneumonia) (Infections and infestations) | 5 | 1
Infection with unknown ANC, Upper airway NOS (Infections and infestations) | 1 | 1
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Device/Prosthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, Extremity - upper (Musculoskeletal and connective tissue disorders) | 0 | 1
Apnea (Nervous system disorders) | 1 | 0
CNS ischemia (Nervous system disorders) | 7 | 1
Confusion (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Neurology - Other (Nervous system disorders) | 1 | 4
Neuropathy: motor (Nervous system disorders) | 0 | 5
Neuropathy: sensory (Nervous system disorders) | 1 | 1
Pyramidal tract dysfunction (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0
Speech impairment (Nervous system disorders) | 1 | 0
Syncope (Fainting) (Nervous system disorders) | 0 | 1
Renal - Other (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chest tube drainage or leak (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 35 | 30
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
CNS hemorrhage (Vascular disorders) | 1 | 0
Hemorrhage pulmonary, Bronchopulmonary NOS (Vascular disorders) | 1 | 0
Hemorrhage pulmonary, Lung (Vascular disorders) | 1 | 0
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 1 | 0
Hemorrhage, GI, Rectum (Vascular disorders) | 0 | 1
Thrombosis/Embolism (vascular access) (Vascular disorders) | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 5 | 6
Vascular - Other (Vascular disorders) | 1 | 0
Pain, Head/Headache (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=346) | Placebo (N=351)
Hemoglobin (Blood and lymphatic system disorders) | 24 | 17
Hypertension (Cardiac disorders) | 68 | 16
Anorexia (Gastrointestinal disorders) | 104 | 61
Constipation (Gastrointestinal disorders) | 49 | 48
Diarrhea (Gastrointestinal disorders) | 123 | 42
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 58 | 15
Nausea (Gastrointestinal disorders) | 58 | 56
Vomiting (Gastrointestinal disorders) | 51 | 44
Fatigue (General disorders) | 125 | 97
Fever (General disorders) | 39 | 18
Insomnia (General disorders) | 30 | 20
Pain, Abdomen NOS (General disorders) | 34 | 12
Pain, Back (General disorders) | 33 | 37
Pain, Bone (General disorders) | 19 | 28
Pain, Chest wall (General disorders) | 23 | 18
Pain, Chest/Thorax NOS (General disorders) | 44 | 32
Pain, Extremity - limb (General disorders) | 25 | 20
Pain, Head/Headache (General disorders) | 38 | 26
Pain, Joint (General disorders) | 30 | 22
Pain, Muscle (General disorders) | 18 | 14
Weight loss (General disorders) | 43 | 17
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 15 | 19
ALT (Metabolism and nutrition disorders) | 26 | 10
AST (Metabolism and nutrition disorders) | 24 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 9
Hypokalemia (Metabolism and nutrition disorders) | 24 | 3
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 18 | 4
Proteinuria (Metabolism and nutrition disorders) | 27 | 6
Dizziness (Nervous system disorders) | 20 | 12
Neuropathy: sensory (Nervous system disorders) | 18 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 67
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 83 | 86
Voice changes (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 65 | 4
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 190 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 15
Rash/desquamation (Skin and subcutaneous tissue disorders) | 140 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must discuss and obtain written consent of the sponsor on the intended publication. The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of the submission in order to obtain approval.